CLINICAL TRIAL: NCT05571852
Title: Before-and-after Study on the Impact of a Home-based Personalized Computerized Training Program on Cognitive Dysfunction Associated With Long COVID
Brief Title: Personalized Computerized Training Program for Cognitive Dysfunction After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Antonio de Nebrija (Other)
Responsible Party: Principal Investigator, Jon Andoni Duñabeitia, Principal Investigator, Universidad Antonio de Nebrija
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UANebrija
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Post-Acute COVID-19; Long COVID
Keywords: Long COVID; Computerized Cognitive Training; Post-Acute Sequeale of COVID-19; Cognitive Dysfunction; Brain Fog
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Cognitive Dysfunction; Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized Cognitive Training (Experimental): Participants will be asked to complete short sessions of around 10 minutes each consisting of a variety of games designed to train the five cognitive skills (attention, memory, coordination, reasoning and perception). Each training session include two games selected among a pool of 12 different games. Participants will be asked to complete a training lasting for 8 weeks in which they could access the training platform as frequently as they wanted.
  Interventions: Device: CogniFit's CCT Post COVID-19

INTERVENTIONS:
Device: CogniFit's CCT Post COVID-19 — The computerized cognitive training (CCT) program is tailored to each person's specific cognitive strengths and weaknesses detected in the Cognitive Assessment Battery (CAB)™ PRO (CogniFit Inc., San Francisco, US; https://www.cognifit.com/cab) by a patented Individualized Training System™ (ITS) software.

SUMMARY:
This before-and-after study aims to evaluate the usefulness and efficacy of a personalized computerized cognitive training (CCT) to improve cognitive function among people with post-acute sequelae of COVID-19 (PASC).

DETAILED DESCRIPTION:
Through an online platform created for the study, adults who self-reported cognitive impairment more than 3 months after receiving a COVID-19 diagnosis will be enlisted and their cognitive status will be assessed using a commercially available test. After determining their level of general cognitive dysfunction, those who qualify and meet the inclusion criteria will be invited to use a customized computerized cognitive training (CCT) program at home and to complete as many daily training sessions as they would want over the course of eight weeks. The sessions will consist of gamified cognitively demanding exercises that target five cognitive skills: attention, coordination, memory, perception, and reasoning. Participants will also complete the general cognitive function assessment at the end of the intervention period, and the differences between the cognitive scores obtained before and after this period will be used as the main outcome measure. Additional analysis will be performed to better characterize the impact of the CCT by exploring the role of the age of the participants, their self-perceive health at baseline, the intensity of the training and the time from initial COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults (older than 18 years old).
* History of infection with COVID-19 at least 3 months prior to expression of interest.
* Presence of self-perceived cognitive dysfunction associated with PACS (concentration problems or brain fog).

Exclusion Criteria:

* Completion of less than 10 training sessions.
* Not completing the final evaluation after the 8-week training period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Cognitive Gains | 8 weeks
  The difference in scores between the initial and final assessments as evaluated by the Cognitive Assessment Battery (CAB)™ PRO

SECONDARY OUTCOMES:
Intensity of the training | 8 weeks
  Number of minutes dedicated to the CCT

CONTACTS AND LOCATIONS:
Overall Officials: Jon Andoni Duñabeitia, Principal Investigator — Universidad Nebrija
Locations (1):
- Universidad Nebrija, Madrid, Spain

REFERENCES:
- [Derived] Dunabeitia JA, Mera F, Baro O, Jadad-Garcia T, Jadad AR. Personalized Computerized Training for Cognitive Dysfunction after COVID-19: A Before-and-After Feasibility Pilot Study. Int J Environ Res Public Health. 2023 Feb 10;20(4):3100. doi: 10.3390/ijerph20043100. PMID 36833793